CLINICAL TRIAL: NCT00864591
Title: Stress Adenosine Cardiac MR Comparison With SPECT Imaging
Brief Title: Stress Adenosine Cardiac Magnetic Resonance (MR) Comparison With Single Photon Emission Computed Tomography (SPECT) Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Orly Goitein MD, Sheba Medical Center
Other Study IDs: SHEBA-08-5654-OG-CTIL
Record Dates: First submitted 2009-03-04; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease; Cardiac Perfusion
Keywords: SPECT Imaging; Stress adenosine CMR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SPECT and stress CMR patients: patients undergoing SPECT stress imaging, for the evaluation of myocardial ischemia.
  The study group will include patients with either normal undergoing SPECT stress imaging or with mild to severe ischemia, to include the entire spectrum of coronary artery disease.
  Patients will be pre selected and evaluated by a non-dependent cardiologist in order to verify that patients in whom the repeat stress might pose a serious risk will be excluded from the study.
  Interventions: Procedure: SPECT Imaging; Procedure: Stress Adenosine CMR

INTERVENTIONS:
Procedure: SPECT Imaging — Myocardial SPECT imaging will be performed 10-12 minutes after the stress injection of Tl-201, at 4 hours, and at 18-24 hours in patients with non-reversible or partially reversible defect on 4-hour imaging. Images will be obtained with a rotating single- or dual-head gamma camera equipped with low-energy high resolution collimators. Energy windows of 20% and 10% will be centered on the 70 KeV and 167 KeV peaks of Tl-201, respectively. Thirty images will be obtained (40 seconds each for the stress and 4-hour redistribution imaging, and 60 seconds each for the 18-24-hour imaging) over 180° extending from the 45° right anterior oblique to the 45° left posterior oblique projections.Localization of the disease in the left anterior descending artery (LAD), left circumflex (Cx) and right coronary artery (RCA) will be performed using a quantitative analysis software.
Procedure: Stress Adenosine CMR — CMR will be performed using a 3-T scanner and a dedicated eight-element cardiac phased-array coil Cine CMR will be performed using steady state free precession in the short-axis, two chamber, three chamber and four-chamber, 8 mm thick, separated by 0-mm gaps.
  Adenosine perfusion CMR: Adenosine will be administered intravenously at 140 µg/kg/min over 6 min. Four minutes into the infusion (or earlier if angina is provoked), a bolus (0.1 mmol/kg at 5 ml/s) of Gadolinium DTPA will be administered. Patients will be instructed to hold their breath. Stress perfusion images will be acquired in the short axis plane (parameters and planning will be similar for stress and rest perfusion evaluation). The patients will be monitored by vector ECG, noninvasive sphygmomanometry, pulse oximetry and capnography.

SUMMARY:
This study is designed to determine the diagnostic value of adenosine cardiac magnetic resonance (CMR) when compared with SPECT.

The investigators hypothesized that adenosine CMR could detect ischemia and is not inferior to SPECT imaging. In addition stress adenosine cardiac MRI offers a "one stop shop" enabling evaluation of cardiac function, rest and stress perfusion and viability.

ELIGIBILITY:
Inclusion Criteria:

* Suspected ischemia referred to SPECT stress imaging

Exclusion Criteria:

* Standard contraindications to MRI including (pacemaker/defibrillator, metallic clips on brain aneurysms, metal fragment in the eye, etc...)
* Congestive heart failure.
* Hemodynamic instability.
* History of asthma or bronchospastic disease.
* Arrhythmia
* Creatinine >1.4
* Non compliant patient, not able to lie supine in the MRI scanner for 1 hour.
* Pregnant patients
* Patients for whom the repeat stress might pose a significant risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing SPECT stress imaging, for the evaluation of myocardial ischemia.
  The study group will include patients with either normal undergoing SPECT stress imaging or with mild to severe ischemia, to include the entire spectrum of coronary artery disease.
  Patients will be pre selected and evaluated by a non-dependent cardiologist in order to verify that patients in whom the repeat stress might pose a serious risk will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Stress adenosine cardiac MRIis not inferior to SPECT imaging in diagnosing myocardial ischemia | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel